CLINICAL TRIAL: NCT00123747
Title: A Phase II Study of 18F-Fluorodeoxyglucose (FluGlucoScan) in Patients Receiving a Treatment Planning Study of 3 Dimensional Conformal Radiation Therapy Guided by Breath Held CT and PET Imaging for Patients With Non-Small Cell Lung Cancer
Brief Title: Study of 18F-Fluorodeoxyglucose (FluGlucoScan) in Patients Receiving a Treatment Planning Study of 3 Dimensional Conformal Radiation Therapy Guided by Breath Held CT and PET Imaging for Patients With Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: Cross Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LU-11-0044/DX-FDG-007/21389
Record Dates: First submitted 2005-07-22; First posted 2005-07-26 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2012-03

CONDITIONS: Lung Neoplasms
Keywords: Positron Emission Tomography; Fluorodeoxyglucose F18; Tomography scanners, X-Ray Computed
MeSH Terms: conditions — Lung Neoplasms | interventions — Magnetic Resonance Spectroscopy; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Positron Emission Tomography (PET) scan Imaging

SUMMARY:
At this time, computed tomography (CT) is the standard tool used at this institution for the staging of non-small cell lung cancer (NSCLC). For most patients, treatment planning for NSCLC is performed with the patient breathing freely during CT scanning. However, recent research has demonstrated that, by holding one's breath briefly, the NSCLC tumor mass can be held motionless. As a result, the tissue to be treated is better pinpointed and the area treated is significantly decreased through breath-hold planning. This allows for a higher dose of radiation to be given to the cancer. PET scanning is a promising newer imaging modality which has shown to be useful in staging NSCLC. This study hypothesizes that breath-held PET scanning and breath held-CT scanning will allow for more stringent radiotherapy plans, minimizing normal tissue toxicity, as well as potentially increasing the dose deliverable to the primary tumor.

DETAILED DESCRIPTION:
Concurrent chemotherapy and 3-dimensional conformal radiation therapy (3D-CRT), using computed-tomography (CT) simulation, is the current standard approach in the treatment of inoperable non-small-cell lung cancer (NSCLC). Despite such therapeutic benefit, local recurrence nonetheless remains a significant impediment to cure. Attempts to improve the accuracy of CT-scanning in radiotherapy treatment planning have been increasingly studied. One such approach is the attempted correlation of CT imaging temporally with the physiologic breathing cycle, a process known as gating. By imaging the tumor only when the tumor is immobilized, gating effectively eliminates the effect of motion, thus leading to typically smaller visible tumor masses and the loss of motion-induced distortions. Lung-tumor immobilization using self-gated breath-holding at extremes of inspiration has been validated clinically, and is associated with improved lung-outcome predictors and normal tissue complication probability overall. Several recent studies have demonstrated PET to be both highly sensitive and moderately to highly specific in the staging of NSCLC, and even more sensitive and specific than CT-scanning in the detection of mediastinal and distant metastases from NSCLC. The co-registration of CT and PET images enables even greater accuracy than either modality alone, while the functional imaging inherent in PET may better facilitate the distinction between benign and malignant structures. Overall, the superior tumor staging capability of PET (or PET-CT fusion) together with the improved dosimetry & diminished normal-tissue toxicity associated with deep inspiration breath-hold (DIBH) is expected to confer considerable clinical advantage to the use of gated PET in the radiotherapeutic planning and treatment of NSCLC.

The first objective is to define the effect of respiratory-gating on PET-based radiotherapy planning in comparison to the free-breathing condition for patients with NSCLC. The endpoints here will be to quantify the variation of both PTV and normal-tissue complication probability (NTCP) for certain relevant organs (lung, esophagus, heart) via a direct analysis of calculated volumes.

The second objective is to identify the correlation between PET-based radiotherapy planning volumes and CT-based planning volumes for respiratory-gated patients with NSCLC. The endpoint for this objective will be to quantify the breath-held, PET-based PTVs and NTCPs in comparison to the breath-held, CT-based PTVs and NTCPs.

This study will consider patients with locally advanced non-small-cell cancer of the lung (NSCLC) who are eligible for radical (i.e. with curative intent) combined-modality therapy. Patients will be accrued from the new patient lung clinic at the Cross Cancer Institute. Following a complete clinical assessment comprising a thorough history and physical examination, a thorough analysis of all available imaging, a consideration of all available laboratory results and consideration of any ancillary test results (e.g. pulmonary function testing), a decision will be made whether or not to offer a patient radical therapy. In the case of any uncertainties, further tests, such as repeat CT scanning or diagnostic PET scanning may be arranged to define eligibility.

Eligibility Criteria:

* Histologically-proven, unresected lung cancer of the following histologic types: *squamous cell carcinoma, *adenocarcinoma, *undifferentiated large cell carcinoma, *non-small cell, not otherwise specified (NOS, diagnosis on cytology alone)
* AJC Stage I-III disease (if all detectable tumor can be encompassed by radiation therapy fields, including both the primary tumor and the involved regional lymph nodes); patients with positive supraclavicular nodes (N3) are not eligible.
* Age > 18 and Karnofsky performance status > 70
* Measurable disease on the CT and PET images
* Patient must be deemed eligible for radical combined-modality therapy
* All patients must sign a study-specific informed consent form.

Ineligibility Criteria:

* M1 disease
* Karnofsky performance status < 70 and age < 18
* Patients who have undergone complete tumor resection
* Patients with post-resection intrathoracic tumor recurrence
* Evidence of small cell histology
* Prior or concurrent malignancy except non-melanomatous skin cancer (unless disease-free for at least 5 years)
* Prior radiotherapy to the thorax or neck
* Prior chemotherapy
* Patients with myocardial infarction within the preceding 6 months or symptomatic heart disease, including angina, congestive heart failure and uncontrolled arrhythmias
* Pregnant women; patients with childbearing potential must practice appropriate contraception.
* Inability to maintain a state of deep inspiratory breath-hold for a minimum length of time

Statistical Analysis: In a previous study comparing DIBH-gated CT-scanning to free-breathing CT-scanning performed at this institution, it was found that a sample size of 10 patients was appropriate to illustrate both a statistically significant reduction in PTV and a statistically significant reduction in V20 (the volume of lung treated to a dose of =20Gy). For the current study, given that the patient population is essentially the same as the last one, and the fact that PET and CT are comparable imaging modalities for NSCLC in terms of their sensitivity, a total sample size of 10 patients would be an appropriate number to assess the difference between breath-held PET and free-breathing PET (i.e. the first objective). This difference, in terms of both PTV and NTCP, will be assessed for statistical significance with a paired Student's t-test.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Histologically proven, resected lung cancer of the following histologic types:

  * squamous cell carcinoma;
  * adenocarcinoma;
  * undifferentiated large cell carcinoma;
  * non-small cell; and
  * not otherwise specified.
* Age equal to or greater than 18 years
* American Joint Committee (AJC) Stage I-III disease (if all detectable tumours can be encompassed by radiation therapy fields, including both the primary tumour and the involved lymph nodes); patients with positive supraclavicular nodes (N3) are not eligible
* Able and willing to follow instructions and comply with the protocol
* Provide written informed consent prior to participation in this study
* Karnofsky Performance Scale score equal to or greater than 70
* Measurable disease on the CT and PET images
* Patient must be deemed eligible for the radical combined-modality therapy.

Exclusion Criteria:

* Nursing or pregnant females
* MI disease
* N3 disease (patients with positive supraclavicular nodes are not eligible)
* Karnofsky performance status less than 70
* Patients who have undergone complete tumour resection
* Patients with post-resection intrathoracic tumour recurrence
* Evidence of small cell history
* Age less than 18 years
* Prior or concurrent malignancy except non-melanomatous skin cancer (unless disease free for at least 5 years)
* Prior radiotherapy to the thorax or neck
* Prior chemotherapy
* Patients with myocardial infarction within the preceding 6 months or symptomatic heart disease, including angina; congestive heart failure; and uncontrolled arrythmias
* Inability to maintain a state of deep inspiratory breath-hold for a minimum length of time

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2005-08; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
To define the effect of respiratory-gating upon PET based radiotherapeutic treatment planning parameters relative to the free-breathing condition for patients with NSCLC | One year

SECONDARY OUTCOMES:
To define the relationship between PET based treatment planning volumes and CT based treatment planning volumes within the realm of respiratory-gating for patients with NSCLC | One Year

CONTACTS AND LOCATIONS:
Overall Officials: Alexander McEwan, MB, MSc, MD, Principal Investigator — AHS Cancer Control Alberta
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada